CLINICAL TRIAL: NCT03193788
Title: A Prospective Randomized Phase III Trial of Maintenance Pemetrexed Versus Observation in Patients With Recurrent or Metastatic Urothelial Carcinoma Who Completed First Line Platinum-based Chemotherapy Without Disease Progression
Brief Title: Pemetrexed Maintenance in Patients With Urothelial Carcinoma Who Completed First Line Platinum-based Chemotherapy
Acronym: PREMIER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, JLee, Associated Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG GU16-05
Record Dates: First submitted 2016-08-13; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer; Ureter Cancer; Transitional Cell Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ureteral Neoplasms; Carcinoma, Transitional Cell | interventions — Pemetrexed; Folic Acid; Vitamin B 12; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- pemetrexed maintenance (Experimental): Drug: Pemetrexed Maintenance therapy: 500 mg/m^2, IV, on Day 1 of each 21-day cycle until progressive disease or treatment discontinuation.
  Drug: folic acid 1000 μg daily orally from 7 days prior to treatment initiation until the end of treatment
  Drug: vitamin B12 injection 1000 μg IM 7 days prior to treatment initiation and the every then every 3 cycles until the end of treatment
  Drug: dexamethasone 4 mg twice orally for 3 days beginning the day before treatment until the end of treatment
  Interventions: Drug: pemetrexed; Drug: Folic Acid; Drug: Vitamin B12 Injection; Drug: Dexamethasone
- observation (No Intervention): observation group will be observed with best supportive care until progressive disease

INTERVENTIONS:
Drug: pemetrexed — Pemetrexed 500 mg/m2mixed in normal saline 100 mL as a 10 minute IV infusion on day 1 of each 21 day cycle
  Other Names: Alimta
  Arms: pemetrexed maintenance
Drug: Folic Acid — folic acid 1000 μg daily orally from 7 days prior to treatment initiation until the end of treatment
  Other Names: Folvite; FA-8; FaLessa
  Arms: pemetrexed maintenance
Drug: Vitamin B12 Injection — vitamin B12 1000 μg IM 7 days prior to treatment initiation and the end of treatment
  Other Names: Vitabee 12
  Arms: pemetrexed maintenance
Drug: Dexamethasone — Dexamethasone 4 mg twice orally for 3 days beginning the day before treatment until the end of treatment to minimize cutaneous reactions
  Other Names: decadron
  Arms: pemetrexed maintenance

SUMMARY:
This study aims to verify superiority of pemetrexed maintenance to observation for patient without disease progression after 1 st line cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
Patients with unresectable locally advanced, recurrent, or metastatic urothelial carcinoma of bladder, ureter, or renal pelvis who do not experience disease progression after 4 to 6 cycles of 1 st line chemotherapy administration.

After completion of 4-6 cycles, patients without disease progression on CT which is taken within 3 weeks after administration of the last chemotherapy will be randomized within 4 weeks after administration of the last chemotherapy to assign either maintenance group or observation group.

Pemetrexed 500 mg/m 2 mixed in normal saline 100 mL as a 10 minute IV infusion on day 1 of each 21 day cycle, with vitamin supplementation (folic acid 1000μg daily orally from 7 days prior to treatment initiation and vitamin B12 1000 μg IM 7 days prior to treatment initiation and then every 3 cycles). Thereafter, vitamin B12 can be injected on the same day of pemetrexed infusion. Dexamethasone 4 mg orally twice daily for 3 days beginning the day before treatment to minimize cutaneous reactions.

Treatment continues until occurrence of disease progression or intolerable toxicities upto maximum of 16 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmation urothelial cancer of bladder, ureter, or renal pelvis.
2. Patients must present with locally advanced, recurrent or metastatic disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent.
3. Patients who were administered 4-6 cycles of cisplatin-based first line chemotherapy [GP (gemcitabine/cisplatin), classic MVAC (methotrexate/vinblastine/doxorubicin/cisplatin), or dose-dense MVAC] and were planned to undergo regular surveillance
4. ce after confirmation of absence of disease progression on CT taken within 3 week after the administration of the last cycle of 1st line chemotherapy.
5. For patients with recurrent disease who received prior adjuvant or neoadjuvant chemotherapy with cisplatin-containing regimen, the last administration of previous treatment should be administered at least 6 months before start date of 1st line chemotherapy.
6. Measurable disease according RECIST criteria v 1.1.
7. Age 20 years or older
8. ECOG performance status 2 or better
9. Adequate bone marrow, hepatic, and renal function
10. Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

1. Prior systemic chemotherapy or immunotherapy for palliative aim before or after 1st line cisplatin-based chemotherapy. However, prior intravesical chemotherapy or immunotherapy is allowed.
2. Disease progression during or after 1st line cisplatin-based chemotherapy
3. Known CNS metastasis
4. Diagnosis of any serious secondary malignancy within the last 2 years, except for adequately treated basal cell or squamous cell carcinoma of skin, early gastric carcinoma, early stage thyroid carcinoma, insignificant prostate carcinoma, or in situ carcinoma of cervix uteri
5. Pregnancy or breast feeding.
6. Serious hypersensitivity reaction to pemetrexed.
7. Severe renal function impairment with creatinine clearance <45 mL/min by standard Cockcroft-Gault formula or GFR measured by Tc99m-DPTA serum clearance method.
8. Other severe acute or chronic medical or psychiatric condition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival | Every 9 weeks, from date of randomization until the date of first documented progression upto 24 months
  Time between randomization and disease progression or death from any causes, whichever came first. Alive patients free of progression will be censored at the last follow-up

SECONDARY OUTCOMES:
objective response rate | every 9 weeks, assess the best overall response from date of randomization until the date of first documented progression upto 24 months
  Objective response rate will be measured according to RECIST 1.1
Incidence of treatment-emergent adverse events | every 3 weeks for pemetrexed group, every 9 weeks for observation group from date of randomization until the date of first documented progression upto 24 months
  Safety assessed per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03
overall survival | From date of randomization until the date of death from any cause, assessed up to 1 year after the end of treatment
  Time interval between randomization and death (all causes). Alive patients will be censored at the last date of news or data cut off
Quality of Life | before randomization, then 9, 18, and 27 weeks after randomization
  QoL will be assessed by EORTC QLQ-C30 core questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Lyun Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (21):
- South Korea (21):
  - Hallym University Medical Center, Hallym University College of Medicine, Anyang
  - Keimyeong University Dongsan Medical Center, Daegu
  - Fatima Hospital, Daegu
  - Chungnam University Hospital, Daejeon
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Gil Medical Center, Incheon
  - Dong-A University Medical Center, Pusan
  - Inje University Haeundae Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan National University School of Medicine, Pusan
  - Asan Medical Center, Seoul
  - Chung Ang University Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Cancer Research Institute, Seoul National University College of Medicine, Seoul
  - Seoul St. Mary's Hospital, College of Medicine, The Catholic University of Korea, Seoul
  - Yonsei Cancer Center, Seoul
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon
  - Uijeongbu St Mary's hospital, Catholic university of Korea, Uijeongbu-si
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] von der Maase H, Hansen SW, Roberts JT, Dogliotti L, Oliver T, Moore MJ, Bodrogi I, Albers P, Knuth A, Lippert CM, Kerbrat P, Sanchez Rovira P, Wersall P, Cleall SP, Roychowdhury DF, Tomlin I, Visseren-Grul CM, Conte PF. Gemcitabine and cisplatin versus methotrexate, vinblastine, doxorubicin, and cisplatin in advanced or metastatic bladder cancer: results of a large, randomized, multinational, multicenter, phase III study. J Clin Oncol. 2000 Sep;18(17):3068-77. doi: 10.1200/JCO.2000.18.17.3068. PMID 11001674
- [Result] Paz-Ares LG, de Marinis F, Dediu M, Thomas M, Pujol JL, Bidoli P, Molinier O, Sahoo TP, Laack E, Reck M, Corral J, Melemed S, John W, Chouaki N, Zimmermann AH, Visseren-Grul C, Gridelli C. PARAMOUNT: Final overall survival results of the phase III study of maintenance pemetrexed versus placebo immediately after induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. J Clin Oncol. 2013 Aug 10;31(23):2895-902. doi: 10.1200/JCO.2012.47.1102. Epub 2013 Jul 8. PMID 23835707
- [Result] Bellmunt J, Theodore C, Demkov T, Komyakov B, Sengelov L, Daugaard G, Caty A, Carles J, Jagiello-Gruszfeld A, Karyakin O, Delgado FM, Hurteloup P, Winquist E, Morsli N, Salhi Y, Culine S, von der Maase H. Phase III trial of vinflunine plus best supportive care compared with best supportive care alone after a platinum-containing regimen in patients with advanced transitional cell carcinoma of the urothelial tract. J Clin Oncol. 2009 Sep 20;27(27):4454-61. doi: 10.1200/JCO.2008.20.5534. Epub 2009 Aug 17. PMID 19687335
- [Result] Vaughn DJ, Broome CM, Hussain M, Gutheil JC, Markowitz AB. Phase II trial of weekly paclitaxel in patients with previously treated advanced urothelial cancer. J Clin Oncol. 2002 Feb 15;20(4):937-40. doi: 10.1200/JCO.2002.20.4.937. PMID 11844814
- [Result] Sweeney CJ, Roth BJ, Kabbinavar FF, Vaughn DJ, Arning M, Curiel RE, Obasaju CK, Wang Y, Nicol SJ, Kaufman DS. Phase II study of pemetrexed for second-line treatment of transitional cell cancer of the urothelium. J Clin Oncol. 2006 Jul 20;24(21):3451-7. doi: 10.1200/JCO.2005.03.6699. PMID 16849761
- [Result] Galsky MD, Moshier E, Krege S, Lin CC, Hahn N, Ecke T, Sonpavde G, Pond G, Godbold J, Oh WK, Bamias A. Posttreatment prognostic nomogram for patients with metastatic urothelial cancer completing first-line cisplatin-based chemotherapy. Urol Oncol. 2014 Jan;32(1):48.e1-8. doi: 10.1016/j.urolonc.2013.07.001. Epub 2013 Sep 18. PMID 24055428